CLINICAL TRIAL: NCT06055764
Title: Role of FDG PET/CT in Patients With Metastasis of Unknown Origin
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mamdouh, Demonstrator of nuclear medicine Assiut university, Assiut University
Other Study IDs: PET/CT in MUO
Record Dates: First submitted 2023-09-12; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET/CT — Patient preparation: Patients will fast for 4 - 6 h before PET scanning to optimize the blood sugar level to 160mg/dl. F-18 FDG dose was 0.14 mCi/kg and injected via intravenous route. During the uptake phase of 18F-FDG patients will be rested in a quite warm room.
  Procedure:
  All PET-CT studies will be done at the nuclear medicine unit in Assuit University Hospital.
  PET-CT images will be interpreted at a workstation equipped with fusion software that offers multi-planar reformatted images and enables display of the PET images, CT images, and fused PET/CT images.

SUMMARY:
Evaluatation of the role of F18FDG-PET/CT in patients with metastases of unknown origin.

DETAILED DESCRIPTION:
Cancer of unknown primary origin (CUP) includes a cluster of heterogeneous tumors that have exceptional clinical features: it is defined as early apparent metastatic disease with no recognizable primary site at the time of presentation. The incidence of CUP ranges around 2% of all new cancer diagnoses.

The work up list of CUP include; a biopsy proven malignancy, a detailed physical examination, many laboratory, radiological and endoscopy. However, these investigations may be costly time-consuming and may eventually fail to detect the site of the primary malignant tumor in the majority of patients. In this context, positron-emission tomography (PET) combined with computed tomography (PET/CT), using the radiotracer 18F fluoro- 2-deoxyglucose (FDG) is an alternative, non-invasive imaging modality with accurate diagnostic performance. It considered good tool for diagnosis of patients with CUP . The basis for use of FDG as radiotracer for PET imaging in CUP depends on the fact that most of the malignant cancer phenotypes show an increased glucose metabolism rate.

Failure to identify the primary tumor hampers optimization of management planning, which in turn may adversely influence patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age more than 18 years presented with either pathologically proved metastases of unknown primary or
* Patients with clinico-radiological suspicious of having metastases.

Exclusion Criteria:

* • Age below 18 years,

  * patients with pathologically proved primary tumor,
  * Patients suffering from advanced disease and in-cooperative patients.
  * Pregnant and lactating women.
  * Patients who had motion artifacts, or those who can't stay stable or calm during acquisition.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will recruit patients with suspected or proven MUO referred to the nuclear medicine unit to detect primary site.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Role of FDG PET/CT in patients with metastasis of unknown origin. Role of FDG PET/CT in patients with metastasis of unknown origin. | through study completion an average 2 years
  patients with metastasis of unknown origin will do PET/CT searching for primary and find if it will change management or not
  Procedure:
  All PET-CT studies will be done at the nuclear medicine unit in Assuit University Hospital.
  PET-CT images will be interpreted at a workstation equipped with fusion software that offers multi-planar reformatted images and enables display of the PET images, CT images, and fused PET/CT images.

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Mamdouh, Principal Investigator — Assiut University

REFERENCES:
- [Background] Park JS, Yim JJ, Kang WJ, Chung JK, Yoo CG, Kim YW, Han SK, Shim YS, Lee SM. Detection of primary sites in unknown primary tumors using FDG-PET or FDG-PET/CT. BMC Res Notes. 2011 Mar 9;4:56. doi: 10.1186/1756-0500-4-56. PMID 21385465
- [Background] Kwee TC, Kwee RM. Combined FDG-PET/CT for the detection of unknown primary tumors: systematic review and meta-analysis. Eur Radiol. 2009 Mar;19(3):731-44. doi: 10.1007/s00330-008-1194-4. Epub 2008 Oct 17. PMID 18925401